CLINICAL TRIAL: NCT05567172
Title: A Pilot Study to Assess WATCHMAN FLX™ Pro Implants by Cardiac Computed Tomography, Magnetic Resonance Imaging and Transesophageal Echocardiography: WATCHMAN FLX Pro CT
Brief Title: Watchman FLX Pro CT Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2517
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-valvular Atrial Fibrillation (AF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Watchman FLX Pro (Experimental)
  Interventions: Device: Left atrial appendage closure device WM FLX Pro

INTERVENTIONS:
Device: Left atrial appendage closure device WM FLX Pro — Left atrial appendage closure

SUMMARY:
The primary objective of this study is to measure device tissue coverage post-implantation of the WATCHMAN FLX™ Pro Left Atrial Appendage Closure (LAAC) Device (WATCHMAN FLX Pro) using the serial advanced imaging modalities of cardiac computed tomography (CT) and transesophageal echocardiography (TEE) and assess its relationship, if any, to clinical events.

DETAILED DESCRIPTION:
WATCHMAN FLX™ Pro CT is a prospective, single-arm, single-center, premarket investigation to assess device tissue coverage in subjects with non-valvular atrial fibrillation (AF) who receive the WATCHMAN FLX Pro device to reduce the risk of stroke. Serial advanced imaging modalities such as CT and TEE will be used. A core laboratory will independently assess select results.

A subject is considered enrolled in the study when the subject or the subject's legally authorized representative signs an Informed Consent Form (ICF) approved by the Independent Ethics Committee (IEC). Up to 50 subjects in whom placement of a WATCHMAN FLX Pro device is attempted will be enrolled.

A baseline assessment including TEE and/or CT imaging with optional cardiac magnetic resonance imaging (MRI) will be done within 7 days prior to the index procedure following core laboratory guidelines. Follow-up clinical assessment and imaging will occur at 14 days, 45 days, and 3 months post index procedure; only clinical assessment will be required at 12 months (unless an in-person assessment is required based on other data). Subjects who are enrolled but not implanted with a WATCHMAN FLX Pro LAAC device will be followed for safety through 12 months after the initial attempted index procedure but will not undergo imaging assessments or evaluation of biochemical markers including measures of coagulation, platelet and endothelial activation and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is of legal age to participate in the study per the laws of their respective geography.
* Subject has documented non-valvular atrial fibrillation (i.e., atrial fibrillation in the absence of moderate or greater mitral stenosis or a mechanical heart valve).
* Subject is clinically indicated for a WATCHMAN FLX Pro device.
* Subject is deemed suitable for the protocol-defined pharmacologic regimen.
* Subject or legal representative is able to understand and willing to provide written informed consent to participate in the study.
* Subject is able and willing to return for required follow-up visits and examinations.

Exclusion Criteria:

* Exclusion criteria are listed below.
* Subject is currently enrolled in another investigational study, except if the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatment.
* Subject has eGFR <30 mL/min (chronic kidney disease stage IV or stage V).
* Subject is contraindicated for TEE.
* Subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction (e.g., due to an underlying hypercoagulable state).
* Subject had or is planning to have any cardiac or non-cardiac intervention or surgical procedure within 30 days prior to or 60 days after implant (including, but not limited to, cardioversion, percutaneous coronary intervention, cardiac ablation, cataract surgery, etc.).
* Subject had a prior stroke (of any cause, whether ischemic or hemorrhagic) or TIA within the 30 days prior to enrollment.
* Subject had a prior major bleeding event per ISTH definitions within the 30 days prior to enrollment. Lack of resolution of related clinical sequelae or planned and pending interventions to resolve bleeding/bleeding source are a further exclusion regardless of timing of the bleeding event.
* Subject has an active bleed.
* Subject has a reversible cause for AF or has transient AF.
* Subject has no LAA or the LAA is surgically ligated.
* Subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 30 days prior to enrollment.
* Subject has a history of atrial septal repair or has an atrial septal defect/patent foramen ovale (ASD/PFO) device.
* Subject has a known contraindication to percutaneous catheterization procedure.
* Subject has a cardiac tumor.
* Subject has signs/symptoms of acute or chronic pericarditis.
* Subject has an active infection.
* There is evidence of tamponade physiology.
* Subject has New York Heart Association Class IV congestive heart failure at the time of enrollment.
* Subject is of childbearing potential and is, or plans to become, pregnant during the time of the study (method of assessment per study physician's discretion).
* Subject has a documented life expectancy of less than 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Device Arm: Watchman FLX Pro: Left atrial appendage closure device
Period: Overall Study
Arm/Group | Device Arm
Started | 43
Completed | 40
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Device Arm: Watchman FLX Pro Device Implantation
Arm/Group | Device Arm
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Hypoattenuated Thickening (HAT) on the Surface of the Device
Description: Serial measurement of any HAT on the surface of the device at 14 days, 45 days and 3 months post implant as assessed by core lab using CT imaging
Time Frame: 14 days to 3 months post implant
Measure: Count of Participants; unit: Participants
Groups:
- 14 Days: Watchman FLX Pro 14 days post device implantation
- 45 Days: Watchman FLX Pro 45 days post device implantation
- 3 Months: Watchman FLX Pro 3 months post device implantation
Arm/Group | 14 Days | 45 Days | 3 Months
Number analyzed (Participants) | 43 | 39 | 42
Participants | 3 | 5 | 5

ADVERSE EVENTS:
Time Frame: 12 Months
Description: Site Reported
Groups:
- Device Arm: Watchman FLX Pro device implantation: Left atrial appendage closure using the Watchman FLX Pro device
Arm/Group | Device Arm
All-Cause Mortality (participants affected / at risk) | 3/43
Serious Adverse Events (participants affected / at risk) | 23/43
Other Adverse Events (participants affected / at risk) | 9/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Arm (N=43)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Cardiac Failure (Cardiac disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 1 (2)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (4)
Device leakage (Product Issues) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism arterial (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Arm (N=43)
GI bleeding (Gastrointestinal disorders) | 1 (2)
Catheter site bleeding (General disorders) | 3 (3)
Device related thrombosis (General disorders) | 2 (2)
Device leakage (Product Issues) | 2 (2)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Groin hematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05567172/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT05567172/SAP_001.pdf